CLINICAL TRIAL: NCT05832606
Title: Food Intervention to Reduce Immunotherapy ToXicity
Acronym: FORX01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FORX01
Record Dates: First submitted 2023-03-21; First posted 2023-04-27 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-12

CONDITIONS: Immune-related Adverse Event; Dietary Habits
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: The FORX interventional trial will be a monocentric single arm dietary intervention trial in 60 patients starting immune checkpoint inhibitor therapy for different types of cancer in both the adjuvant and metastatic setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- High Fiber diet (Experimental): During the first 12 weeks of immune checkpoint inhibitor therapy, patients will receive weekly boxes containing 30 different plants (vegetables, fruits, nuts, grains) according to seasonal availability following the Flemish Superior Health Council guidelines. Recipes will be added to inspire processing of the box. Boxes will be ordered at an online supermarket, who will deliver the boxes at patients' homes. Weekly follow-up will ensure a minimum daily intake of 20 g of fiber, progressively increasing over the first 4 weeks.
  Interventions: Other: Food box containing 30 different plants

INTERVENTIONS:
Other: Food box containing 30 different plants — Food boxes during first 12 weeks of therapy. Clinical follow-up until end of immunotherapy.

SUMMARY:
The FORX (Food intervention to Reduce immunotherapy toXicity) trial will assess whether supplementing dietary fiber intake by providing weekly boxes containing 30 different plants to patients with solid tumors starting immune checkpoint inhibitor therapy affects the incidence of immune related adverse events.

DETAILED DESCRIPTION:
Immune checkpoint inhibitor (ICI) therapy has revolutionized cancer treatment but can give rise to immune related adverse events (irAEs) that are currently not preventable. These irAEs impact patients' quality of life and oncological treatment course. The gut plays an essential role in immune homeostasis and gut dysbiosis is implicated in (auto)inflammatory conditions. The FORX trial investigates whether the composition of the gut microbiome can be altered to improve ICI tolerance. It has been shown that healthy volunteers who ingest at least 30 different plants (vegetables, fruits, nuts) weekly, have a more diverse microbiome than those who consume 10 or less. A fiber-rich diet has been associated with improved outcome of ICI treatment. This trial is the first prospective trial to translate these findings into a concrete dietary advice. The diets of patients with a solid tumor who start ICI will be supplemented by weekly boxes containing 30 different plants during the first 12 weeks of their treatment. The increased fiber intake is expected to strengthen the gut microbiome and reduce the incidence of irAEs. Stool and blood samples will clarify the microbial and cytokine signatures associated with irAEs. The FORX trial will provide valuable insights in the interaction between the gut microbiome and autoimmunity and serve as a basis for nutritional advice and the development of targeted probiotics. It will empower cancer patients and improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* solid tumor starting anti-programmed cell death protein 1 (anti-PD1) and/or anti-cytotoxic T-lymphocyte-associated antigen 4 (anti-CTLA4) antibodies as part of standard of care.
* able to sign informed consent.

Exclusion Criteria:

* no oral intake possible.
* probiotic use and unwillingness to stop during the trial.
* combination therapy with chemotherapy or targeted agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of performing a dietary intervention trial in our center | 12 weeks
  Recruitment will be temporarily held after 10 patients to assess compliance with protocol and dietary intervention. If at least 7/10 patients are able to complete the 12 weeks according to protocol, the trial will be considered feasible and recruitment will continue.
Incidence of immune related adverse events | up to 24 months
  Assess incidence and grade of irAEs throughout the 12-week intervention phase and until end of ICI treatment by frequency counts and grade. Comparison with historical control.

SECONDARY OUTCOMES:
Response rate | up to 48 weeks
  Measure objective response rate at 12 weeks and progression free survival at week 12, 24 and 48 according to RECIST 1.1. Observational comparison with historical control.
Quality of life | 12 weeks
  Assess change in quality of life following dietary intervention using European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) and Hospital Anxiety and Depression Score (HADS) questionnaire at baseline, at 6 weeks and at 12 weeks.
Changes in gut microbiota | 12 weeks and in case of an irAE up to 48 months
  Assess changes in gut microbiota composition following dietary intervention. Assess microbiota signatures associated with irAEs.
Assess changes in cytokines and immune cell subsets associated with irAEs | 12 weeks and in case of an irAE up to 48 months
  Blood samples will be collected at baseline, every 4 weeks for 12 weeks during the intervention and in case of toxicity. Based on published data, the investigators will primarily focus on Th17-related cytokines (IL-6, IL-17, IL-23, IFN-gamma). PBMC will be analysed using high dimensional flow cytometry, using panels to measure different immune cell subsets (T cells and subtypes, B cells, among which regulatory B cells). Analysis using regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Aspeslagh, MD PhD, Principal Investigator — Vrije Universiteit Brussel (VUB), Universitair Ziekenhuis Brussel (UZ Brussel)
Locations (1):
- UZ Brussel, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No